CLINICAL TRIAL: NCT01197716
Title: Deutsches CPU-Register. Unterstützt Durch Die Deutsche Gesellschaft für Kardiologie.
Brief Title: German Chest Pain Unit (CPU)-Register
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: German CPU-Register
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Chest Pain
Keywords: Chest Pain Unit; Myocardial infarction; Register; Admission to a Chest Pain Unit for any reason
MeSH Terms: conditions — Chest Pain; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Chest Pain Unit (CPU) register is a nationwide scientific investigation, in which data concerning the hospital-stay within the Chest Pain Unit are documented. Furthermore, a Follow-up via telephone is conducted after 3 months.

DETAILED DESCRIPTION:
The aim of a Chest Pain Unit (CPU) is to clarify unclear chest pain quickly and specifically. Present data from Germany, the USA and England prove that the organisation models of a CPU lead beside a drastic reduction of mortality also to a cost reduction as well as a shortening of the average inpatient hospital stays.

Therefore it seems reasonable to assign a minimum standard to CPUs. Although there are internationally already standards for CPUs up to complete certification programmes, it is an explicit wish of the German society for cardiology (DGK) to create an own standard which considers on the national circumstances.

The aim of the CPU register is the internal and external validation of the care quality of CPU including Benchmark reports and risk-adjusted comparisons.

ELIGIBILITY:
Inclusion Criteria:

All patients that are admitted to a Chest Pain Unit are included in this register.

Exclusion Criteria:

Missing informed consent (informed consent can NOT be given in the acute phase of the disease, if consciousness is limited at that time; instead the patient will be asked for his consent at a later point of time, when he is fully conscious).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to a chest pain unit in a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 34470 (Actual)
Dates: Start 2008-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Internal and external validation of the medical care quality in the field of Chest Pain Units | hospital stay
  including benchmark reports and risk adjusted comparisons.

SECONDARY OUTCOMES:
Documentation of CPU complications | up to 30 hours on average
  including mortality, serious but non-fatal complications (e.g. stroke, heavy and moderate bleedings) as well as documentation of the medication at hospital discharge
Documentation of long-term mortality and serious but non-fatal complications | 3 months after discharge
  as well as additional hospital admissions and medication

CONTACTS AND LOCATIONS:
Overall Officials: Harald Darius, MD, Study Chair — Vivantes Clinic Neukölln
Locations (1):
- Bethanien Krankenhaus, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No